CLINICAL TRIAL: NCT00384189
Title: A Comparative Study of Inhaled Ciclesonide Versus Placebo in Children With Asthma
Brief Title: A Comparative Study of Inhaled Ciclesonide Versus Placebo in Children (6-11 Years) With Asthma
Acronym: RAINBOW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Nycomed GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BY9010/M1-209; U1111-1172-2297 (Registry Identifier: WHO)
Record Dates: First submitted 2006-10-04; First posted 2006-10-05 (Estimated); Results first posted 2016-08-16 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; children
MeSH Terms: conditions — Asthma | interventions — ciclesonide; Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ciclesonide 40 µg (Active Comparator): Placebo-matching ciclesonide, inhaled via a metered-dose inhaler (MDI) with 1,1,1,2-hydrofluoroalkane (HFA)-134a as propellant, once daily, in the evening for 2 to 4 weeks in the Baseline period followed by ciclesonide 40 µg, inhaled via a MDI with HFA-134a as propellant, once daily in the evening for 12 weeks. Salbutamol 100 μg/puff was available to be used as rescue medication if needed.
  Interventions: Drug: Ciclesonide; Drug: Placebo; Drug: Salbutamol
- Ciclesonide 80 µg (Active Comparator): Placebo-matching ciclesonide, inhaled via a MDI with HFA-134a as propellant, once daily, in the evening for 2 to 4 weeks in the Baseline period followed by ciclesonide 80 µg, inhaled via a MDI with HFA-134a as propellant, once daily in the evening for 12 weeks. Salbutamol 100 μg/puff was available to be used as rescue medication if needed.
  Interventions: Drug: Ciclesonide; Drug: Placebo; Drug: Salbutamol
- Ciclesonide 160 µg (Active Comparator): Placebo-matching ciclesonide, inhaled via a MDI with HFA-134a as propellant, once daily, in the evening for 2 to 4 weeks in the Baseline period followed by ciclesonide 160 µg, inhaled via a MDI with HFA-134a as propellant, once daily in the evening for 12 weeks. Salbutamol 100 μg/puff was available to be used as rescue medication if needed.
  Interventions: Drug: Ciclesonide; Drug: Placebo; Drug: Salbutamol
- Placebo (Placebo Comparator): Placebo-matching Ciclesonide, inhaled via a MDI with HFA-134a as propellant, once daily in the evening for 2 to 4 week in the Baseline period followed by placebo-matching ciclesonide, inhaled via a MDI with HFA-134a as propellant, once daily in the evening for 12 weeks. Salbutamol 100 μg/puff was available to be used as rescue medication if needed.
  Interventions: Drug: Placebo; Drug: Salbutamol

INTERVENTIONS:
Drug: Ciclesonide — inhaled Ciclesonide
  Arms: Ciclesonide 160 µg; Ciclesonide 40 µg; Ciclesonide 80 µg
Drug: Placebo — Ciclesonide placebo-matching inhaler
Drug: Salbutamol — Salbutamol inhalation powder

SUMMARY:
The purpose of this study is to investigate the efficacy of inhaled ciclesonide at three different dose levels compared with placebo with respect to pulmonary function, asthma symptoms, and use of rescue medication in children aged 6-11 years with asthma. Treatment medication will be administered as follows: ciclesonide or placebo will be inhaled once daily in the evening. The study consists of a baseline period (2 to 4 weeks) and a treatment period (12 weeks). The study provides further data on safety and tolerability of ciclesonide.

DETAILED DESCRIPTION:
The drug being tested is called ciclesonide. This study looked at the safety and efficacy of inhaled ciclesonide in children with asthma. The study enrolled 1080 patients.

Participants were randomly assigned to 1 of 4 treatment groups which were undisclosed to the patient and study doctor during the study:• Ciclesonide 40 µg, 80 µg or 160 µg • Placebo- this is similar to study drug but has no active ingredient. Ciclesonide was inhaled via a metered-dose inhaler (MDI with HFA-134a propellant), with or without spacer, once daily in the evening throughout the study. All participants were asked to document daily AM and PM peak expiratory flow (PEF), daytime and nighttime asthma symptom scores and number of puffs of rescue medicine in an electronic diary. This multi-centre trial was conducted worldwide. The overall time to participate in this study was 20 weeks. Participants made multiple visits to the clinic plus a final visit 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Main Inclusion Criteria:

* History of asthma for at least 6 months
* Ability to show optimal use of MDI, including inhalation technique
* Lung function and reversibility within specified limits

Main Exclusion Criteria:

* Concomitant severe diseases
* Diseases which are contraindications for the use of inhaled steroids
* Two or more inpatient hospitalizations for asthma within the last year
* Respiratory tract infection or asthma exacerbation within the last 30 days prior to entry into the study
* Use of systemic steroids within the last 30 days prior to inclusion (depot steroids 6 weeks)
* Beginning of or change in immunotherapy within the last 6 months prior to inclusion
* Inability to follow the procedures of the study

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1080 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (85):
- Bulgaria (4):
  - Altana Pharma/Nycomed, Plovdiv
  - Altana Pharma/Nycomed, Rousse
  - Altana Pharma/Nycomed, Sofia
  - Altana Pharma/Nycomed, Vama
- Germany (13):
  - Altana Pharma/Nycomed, Dresden
  - Altana Pharma/Nycomed, Freising
  - Altana Pharma/Nycomed, Fulda
  - Altana Pharma/Nycomed, Homburg
  - Altana Pharma/Nycomed, Kassel
  - Altana Pharma/Nycomed, Leipzig
  - Altana Pharma/Nycomed, Mannheim
  - Altana Pharma/Nycomed, Marburg
  - Altana Pharma/Nycomed, München
  - Altana Pharma/Nycomed, Rosenheim
  - Altana Pharma/Nycomed, Schwäbisch Hall
  - Altana Pharma/Nycomed, Welzheim
  - Altana Pharma/Nycomed, Wesel
- Hungary (9):
  - Altana Pharma/Nycomed, Budapest
  - Altana Pharma/Nycomed, Debrecen
  - Altana Pharma/Nycomed, Jászberény
  - Altana Pharma/Nycomed, Kiskunhalas
  - Altana Pharma/Nycomed, Miskolc
  - Altana Pharma/Nycomed, Mosdós
  - Altana Pharma/Nycomed, Mosonmagyaróvár
  - Altana Pharma/Nycomed, Pécs
  - Altana Pharma/Nycomed, Szeged
- Poland (7):
  - Altana Pharma/Nycomed, Inowrocław
  - Altana Pharma/Nycomed, Lodz
  - Altana Pharma/Nycomed, Lublin
  - Altana Pharma/Nycomed, Poznan
  - Altana Pharma/Nycomed, Torun
  - Altana Pharma/Nycomed, Warsaw
  - Altana Pharma/Nycomed, Zawadzkie
- Romania (7):
  - Altana Pharma/Nycomed, Brasov
  - Altana Pharma/Nycomed, Bucharest
  - Altana Pharma/Nycomed, Cluj-Napoca
  - Altana Pharma/Nycomed, Craiova
  - Altana Pharma/Nycomed, Galati
  - Altana Pharma/Nycomed, Iași
  - Altana Pharma/Nycomed, Sibiu
- Russia (13):
  - Altana Pharma/Nycomed, Chelyabinsk
  - Altana Pharma/Nycomed, Ivanovo
  - Altana Pharma/Nycomed, Kislovodsk
  - Altana Pharma/Nycomed, Moscow
  - Altana Pharma/Nycomed, Murmansk
  - Altana Pharma/Nycomed, Novosibirsk
  - Altana Pharma/Nycomed, Rostov
  - Altana Pharma/Nycomed, Saint Petersburg
  - Altana Pharma/Nycomed, Samara
  - Altana Pharma/Nycomed, Smolensk
  - Altana Pharma/Nycomed, Tomsk
  - Altana Pharma/Nycomed, Vladimir
  - Altana Pharma/Nycomed, Voronezh
- South Africa (14):
  - Altana Pharma/Nycomed, Bellville - Cape Town -
  - Altana Pharma/Nycomed, Bloemfontein
  - Altana Pharma/Nycomed, Cape Town
  - Altana Pharma/Nycomed, Centurion
  - Altana Pharma/Nycomed, Durban
  - Altana Pharma/Nycomed, Durban, Amanzimtoti
  - Altana Pharma/Nycomed, Gezina, Pretoria
  - Altana Pharma/Nycomed, Morningside, Sandton
  - Altana Pharma/Nycomed, Mowbray, Cape Town
  - Altana Pharma/Nycomed, New Redruth, Alberton
  - Altana Pharma/Nycomed, Panorama / RSA-Cape Town
  - Altana Pharma/Nycomed, Somerset West
  - Altana Pharma/Nycomed, Westville
  - Altana Pharma/Nycomed, Wynberg
- Spain (7):
  - Altana Pharma/Nycomed, Barcelona
  - Altana Pharma/Nycomed, Esplugues de Llobregat
  - Altana Pharma/Nycomed, Leganés
  - Altana Pharma/Nycomed, Madrid
  - Altana Pharma/Nycomed, Manresa
  - Altana Pharma/Nycomed, Sabadell (Barcelona)
  - Altana Pharma/Nycomed, Tarrasa
- Ukraine (11):
  - Altana Pharma/Nycomed, Dnipropetrovsk
  - Altana Pharma/Nycomed, Donetsk
  - Altana Pharma/Nycomed, Kharkiv
  - Altana Pharma/Nycomed, Kiev
  - Altana Pharma/Nycomed, Kyiv
  - Altana Pharma/Nycomed, Lviv
  - Altana Pharma/Nycomed, Odesa
  - Altana Pharma/Nycomed, Poltava
  - Altana Pharma/Nycomed, Simferopol
  - Altana Pharma/Nycomed, Vinnytsia
  - Altana Pharma/Nycomed, Zaporizhzhya

REFERENCES:
- [Derived] Pedersen S, Potter P, Dachev S, Bosheva M, Kaczmarek J, Springer E, Dunkel J, Engelstatter R. Efficacy and safety of three ciclesonide doses vs placebo in children with asthma: the RAINBOW study. Respir Med. 2010 Nov;104(11):1618-28. doi: 10.1016/j.rmed.2010.06.012. Epub 2010 Jul 8. PMID 20619624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 110 investigative sites in Bulgaria, Germany, Hungary, Poland, Romania, Russia, South Africa, Spain, and Ukraine from 29 September 2006 to 17 August 2007.
Pre-assignment Details: Children with a diagnosis of asthma were enrolled equally in 1 of 4 treatment groups, once a day placebo, 40 µg, 80 µg or 160 µg ciclesonide.
Period: Overall Study
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Started | 305 | 312 | 313 | 150
Randomized, Not Treated | 1 | 0 | 2 | 4
Actual Treatment Received | 305 (1 participant randomized to 160 μg who actually received 40 μg is included.) | 312 | 310 (1 participants in the 160 μg arm actually received 40 μg and is moved to that arm.) | 146
Completed | 255 | 255 | 255 | 110
Not Completed | 50 | 57 | 58 | 40
Not completed — Reason Not Specified | 50 | 57 | 58 | 40

BASELINE CHARACTERISTICS:
Population: Full Analysis Set includes all randomized participants who received at least one dose of study drug, as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo | Total
Number analyzed (Participants) | 305 | 312 | 310 | 146 | 1073
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (1.7) | 8.4 (1.6) | 8.7 (1.6) | 8.4 (1.7) | 8.4 (1.6)
Gender [Count of Participants; unit: Participants]
  Female | 95 | 121 | 92 | 54 | 362
  Male | 210 | 191 | 218 | 92 | 711
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 276 | 279 | 277 | 133 | 965
  non-Caucasian | 29 | 33 | 33 | 13 | 108
Region of Enrollment [Number; unit: participants]
  Bulgaria | 29 | 33 | 33 | 15 | 110
  Germany | 17 | 16 | 12 | 8 | 53
  Hungary | 42 | 45 | 43 | 22 | 152
  Poland | 49 | 48 | 49 | 23 | 169
  Romania | 15 | 16 | 21 | 8 | 60
  Russian Federation | 54 | 52 | 55 | 27 | 188
  South Africa | 32 | 34 | 32 | 13 | 111
  Spain | 18 | 18 | 17 | 8 | 61
  Ukraine | 49 | 50 | 48 | 22 | 169
Height [Mean (Standard Deviation); unit: cm] | 134.6 (10.8) | 134.5 (11.0) | 135.9 (10.8) | 134.6 (11.1) | 134.9 (10.9)
Weight [Mean (Standard Deviation); unit: kg] | 32.3 (9.1) | 31.9 (9.3) | 33.2 (9.5) | 32.7 (9.7) | 32.5 (9.4)
Duration of Asthma [Mean (Standard Deviation); unit: months] | 44.3 (27.7) | 45.5 (27.8) | 45.5 (27.4) | 47.6 (28.0) | 45.5 (27.7)
Inhaled Glucocorticosteroids (ICS) Pretreatment [Number; unit: participants]
  Yes | 200 | 204 | 199 | 102 | 705
  No | 105 | 108 | 111 | 44 | 368
ICS Pretreatment Dose [Mean (Standard Deviation); unit: µg/day] — The number of participants with ICS pretreatment dose data is 200, 204, 199 and 102 in each treatment arm, respectively.
  µg/day | 211.9 (181.9) | 222.8 (188.8) | 205.0 (177.1) | 224.6 (178.8) | 214.8 (182.1)
Asthma Severity According to Global Initiative for Asthma (GINA) [Number; unit: participants]
  Intermittent | 20 | 19 | 13 | 7 | 59
  Mild | 25 | 22 | 29 | 10 | 86
  Moderate | 112 | 110 | 104 | 50 | 376
  Severe | 148 | 161 | 164 | 79 | 552

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Peak Expiratory Flow (PEF)
Description: PEF is the maximum speed of expiration. A portable electronic PEF meter was used for the home PEF readings. The patients recorded PEF daily, in the morning immediately after getting up. Readings were done preferably at least 4 hours after use of rescue medication and before inhalation of the study medication. At each measurement, three readings were obtained in the standing position. All three values were recorded in the diary; the highest value was used for evaluation. The higher change from Baseline values are the best. Analysis of covariance (ANCOVA) model with the baseline value and age as covariates was used for analysis. Last observation carried forward.
Time Frame: Baseline and Week 12
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug based on the study drug they were randomized to receive, with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 304 | 312 | 311 | 146
liters/minute | 15.23 (2.69) | 14.79 (2.60) | 17.37 (2.68) | 5.40 (3.71)
Statistical Analysis 1: Comparison: Ciclesonide 40 µg vs Placebo; Test type: Superiority or Other; p = 0.0116, ANCOVA; Baseline value and age as covariates. One-sided p-value, significance level 2.5%; Least Squares Mean Difference = 9.8, 95% CI 2-sided [1.4 to 18.3], Standard Error of Mean 4.3
Statistical Analysis 2: Comparison: Ciclesonide 80 µg vs Placebo; Test type: Superiority or Other; p = 0.0148, ANCOVA; Baseline value and age as covariates. One-sided p-value, significance level 2.5%; Least Square Means Difference = 9.4, 95% CI 2-sided [0.9 to 17.8], Standard Error of Mean 4.3
Statistical Analysis 3: Comparison: Ciclesonide 160 µg vs Placebo; Test type: Superiority or Other; p = 0.0028, ANCOVA; Baseline value and age as covariates. One-sided p-value, significance level 2.5%; Least Squares Means Difference = 12.0, 95% CI 2-sided [3.5 to 20.4], Standard Error of Mean 4.3

2. Secondary Outcome: Time to First Event of Lack of Efficacy (LOE) by Week 12
Description: Kaplan Meier Estimates of the probability of not experiencing LOE by Week 12 was measured. LOE was reached if any of the following criteria occurred during the treatment period: • asthma exacerbation (a worsening of asthma symptoms requiring a change in medication; • nocturnal awakenings due to asthma on any 4 or more nights during any 7-consecutive-day period; • use of more than 8 puffs/day of salbutamol on any 4 or more days during any 7-consecutive-day period; • decrease in morning PEF to <80% of randomization value on any 4 consecutive days during the treatment period.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Percent
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 304 | 312 | 311 | 146
Percent | 72.8 | 74.5 | 73.2 | 66.9
Statistical Analysis 1: Comparison: Ciclesonide 40 µg vs Placebo; Test type: Superiority or Other; p = 0.1362, Log Rank — Two-sided p-value, significance level 5%
Statistical Analysis 2: Comparison: Ciclesonide 80 µg vs Placebo; Test type: Superiority or Other; p = 0.0891, Log Rank — Two-sided p-value, significance level 5%
Statistical Analysis 3: Comparison: Ciclesonide 160 µg vs Placebo; Test type: Superiority or Other; p = 0.1574, Log Rank — Two-sided p-value, significance level 5%

3. Secondary Outcome: Percentage of Days With Asthma Control Based on Symptoms, Use of Rescue Medication, Morning PEF and PEF Fluctuation
Description: Control of asthma was evaluated on a daily basis (24 hours) using the following variables: asthma symptoms, use of rescue medication, morning (am) PEF and PEF fluctuation. The median percentage of days with asthma control is presented.
Time Frame: 28 days prior to last visit (Up to 12 Weeks)
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 302 | 311 | 309 | 144
percentage of days | 7.14 [0.0 to 100.0] | 10.53 [0.0 to 100.0] | 6.67 [0.0 to 100.0] | 0.0 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Ciclesonide 40 µg vs Placebo; Test type: Superiority or Other; p = 0.0010, Wilcoxon (Mann-Whitney) — One-sided p-value for superiority, significance level 2.5%
Statistical Analysis 2: Comparison: Ciclesonide 80 µg vs Placebo; Test type: Superiority or Other; p = 0.0006, Wilcoxon (Mann-Whitney) — One-sided p-value for superiority, significance level 2.5%
Statistical Analysis 3: Comparison: Ciclesonide 160 µg vs Placebo; Test type: Superiority or Other; p = 0.0002, Wilcoxon (Mann-Whitney) — One-sided p-value for superiority, significance level 2.5%

4. Secondary Outcome: Change From Baseline in Lung Function Variable Forced Expiratory Volume in One Second (FEV1)
Description: Spirometry was performed according to local standards. FEV1 is the maximal amount of air forcefully exhaled from the lungs in one second. Higher change numbers indicate better lung function.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 270 | 281 | 270 | 124
liters | 0.123 (0.015) | 0.122 (0.015) | 0.139 (0.015) | 0.039 (0.022)

5. Secondary Outcome: Change From Baseline in Lung Function Variable PEF by Spirometry
Description: Spirometry was performed according to local standards. PEF is the maximum speed of expiration. Analysis was ANCOVA with factors value at Baseline, treatment, age, sex, center pool, ICS pretreatment, spacer use and asthma severity. Higher change numbers indicate better lung function.
Time Frame: Baseline and Week 12
Population: Participants from the Intent-to-treat population, all randomized participants who received at least one dose of study drug based on the study drug they were randomized to receive, with data available for analysis. Last Observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 270 | 281 | 272 | 124
liters/minute | 20.68 (2.61) | 21.71 (2.51) | 22.25 (2.61) | 15.13 (3.69)

6. Secondary Outcome: Change From Baseline in Morning PEF From Diary
Description: PEF is the maximum speed of expiration. A portable electronic PEF meter was used for the home PEF readings. The patients recorded PEF daily, in the morning immediately after getting up. Readings were done preferably at least 4 hours after use of rescue medication and before inhalation of the study medication. At each measurement, three readings were obtained in the standing position. All three values were recorded in the diary; the highest value was used for evaluation. The higher change from Baseline values are the best. Analysis of covariance (ANCOVA) model with the Baseline value and age as covariates was used for analysis.
Time Frame: Baseline and Weeks 1 thru 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 304 | 312 | 311 | 146
liters/minute
  Change at Week 1 (n=303,311,310,146) | 11.61 (1.55) | 9.20 (1.50) | 11.54 (1.54) | 4.54 (2.13)
  Change at Week 2 (n=303,311,310,146) | 9.82 (1.89) | 11.95 (1.83) | 12.26 (1.89) | 4.20 (2.61)
  Change at Week 3 (n=304,312,310,146) | 11.36 (2.08) | 11.11 (2.01) | 13.15 (2.07) | 6.74 (2.87)
  Change at Week 4 (n=304,312,310,146) | 13.63 (2.18) | 13.27 (2.12) | 15.60 (2.18) | 6.31 (3.02)
  Change at Week 5 | 14.86 (2.23) | 13.33 (2.16) | 15.39 (2.22) | 9.67 (3.08)
  Change at Week 6 | 13.91 (2.30) | 13.26 (2.23) | 14.71 (2.29) | 7.64 (3.18)
  Change at Week 7 | 14.57 (2.37) | 15.05 (2.30) | 14.14 (2.36) | 6.21 (3.28)
  Change at Week 8 | 14.57 (2.39) | 15.92 (2.31) | 13.63 (2.38) | 7.05 (3.30)
  Change at Week 9 | 15.26 (2.44) | 16.02 (2.36) | 13.23 (2.43) | 7.88 (3.37)
  Change at Week 10 | 16.35 (2.48) | 16.79 (2.40) | 14.59 (2.47) | 7.66 (3.43)
  Change at Week 11 | 16.12 (2.60) | 15.97 (2.52) | 16.24 (2.59) | 6.80 (3.60)
  Change at Week 12 | 15.93 (2.72) | 15.43 (2.64) | 17.59 (2.71) | 6.41 (3.76)

7. Secondary Outcome: Change From Baseline in Evening PEF From Diary
Description: as for outcome 6
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: liters/minute
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 304 | 312 | 310 | 146
liters/minute | 10.16 (2.54) | 9.37 (2.46) | 12.71 (2.53) | 4.02 (3.52)

8. Secondary Outcome: Change From Baseline in Diurnal PEF Fluctuations
Description: PEF is the maximum speed of expiration. A portable electronic PEF meter was used for the home PEF readings. The patients recorded PEF daily, in the morning immediately after getting up. Readings were done preferably at least 4 hours after use of rescue medication and before inhalation of the study medication. At each measurement, three readings were obtained in the standing position. All three values were recorded in the diary; the highest value was used for evaluation. A negative change from Baseline indicates improvement. Analysis of covariance (ANCOVA) model with the Baseline value and age as covariates was used for analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 303 | 312 | 310 | 146
percent change | -0.841 (9.942) | -1.209 (10.686) | -1.192 (11.290) | 0.214 (9.453)

9. Secondary Outcome: Change in Asthma Symptom Total Score
Description: Measurements of both nighttime and daytime asthma symptoms were assessed on a daily basis by the patient in the electronic diary, according to the following scales: Nighttime Asthma Score using a 5 point scale: 0=no asthma symptoms, slept through the night to 4=bad night, awake most of the night because of asthma. Daytime Asthma Score using a 5 point scale: 0=very well, no asthma symptoms to 4=asthma very bad, unable to carry out daily activities as usual. Total possible overall daily score range from 0(best) to 4 (worst). A negative change from Baseline indicated improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 304 | 312 | 311 | 146
score on a scale
  Asthma Total Symptom Score (n=304,312,310,146) | -0.916 (1.265) | -0.983 (1.209) | -0.879 (1.270) | -0.572 (1.483)
  Asthma Daytime Symptom Score (n=304,312,310,146) | -0.529 (0.682) | -0.553 (0.721) | -0.517 (0.662) | -0.354 (0.801)
  Asthma Nighttime Symptom Score | -0.392 (0.775) | -0.435 (0.672) | -0.350 (0.791) | -0.233 (0.858)

10. Secondary Outcome: Change in Use of Rescue Medications
Description: The daily use of rescue medication (salbutamol) was recorded in the electronic diary in the morning and the evening. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: puffs/day
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 304 | 312 | 311 | 146
puffs/day | -0.872 (1.634) | -0.999 (1.523) | -0.886 (1.771) | -0.527 (1.931)

11. Secondary Outcome: Percentage of Days With Asthma Control Based on Symptoms, Use of Rescue Medication and Morning PEF
Description: Control of asthma was evaluated on a daily basis (24 hours) using the following variables: asthma symptoms, use of rescue medication, and morning (am) PEF. The median percentage of days with asthma control is presented.
Time Frame: 28 days prior to last visit (Up to 12 Weeks)
Population: as for outcome 1
Measure: Median (Full Range); unit: percentage of days
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 302 | 311 | 309 | 144
percentage of days | 8.33 [0.0 to 100.0] | 13.64 [0.0 to 100.0] | 13.04 [0.0 to 100.0] | 0.0 [0.0 to 100.0]

12. Secondary Outcome: Change From Baseline in Pediatric Asthma Quality of Life Questionnaire Standard [PAQLQ(S)] Overall Score
Description: PAQLQS is a disease specific instrument to assess the impact of asthma on the patient's quality of life. The PAQLQS consists of 23 items in 3 domains evaluating activity limitations, symptoms and emotional function. Patients answered each question using a 7-point scale from 1= maximum impairment to 7=no impairment) about their experience during the previous week. Total possible score ranging from 23 (worst) to 161(best). Higher change from Baseline scores are the best. Analysis of covariance (ANCOVA) model with the baseline value and age as covariates was used for analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 167 | 179 | 171 | 76
score on a scale | 0.78 (0.07) | 0.71 (0.07) | 0.72 (0.07) | 0.43 (0.10)

13. Secondary Outcome: Change From Baseline in Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) Overall
Description: PACQLQ assesses the impact of the child's asthma on the quality of life of the caregiver. The PACQLQ consists of 13 items in 2 domains evaluating activity limitations and emotional function. Caregivers answered each question using a 7-point scale from 1= maximum impairment to 7=no impairment about their experience during the previous week. Total possible score ranging from 13 (worst) to 91(best). Higher change from Baseline scores are the best. Analysis of covariance (ANCOVA) model with the baseline value and age as covariates was used for analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Number analyzed (Participants) | 169 | 177 | 172 | 74
score on a scale | 0.82 (0.08) | 0.88 (0.08) | 0.84 (0.08) | 0.71 (0.12)

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days after last dose of study drug (Up to 20 Weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ciclesonide 40 µg | Ciclesonide 80 µg | Ciclesonide 160 µg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/305 | 5/312 | 2/310 | 1/146
Other Adverse Events (participants affected / at risk) | 49/305 | 45/312 | 45/310 | 14/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciclesonide 40 µg (N=305) | Ciclesonide 80 µg (N=312) | Ciclesonide 160 µg (N=310) | Placebo (N=146)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 0
Tonsillitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ciclesonide 40 µg (N=305) | Ciclesonide 80 µg (N=312) | Ciclesonide 160 µg (N=310) | Placebo (N=146)
Nasopharyngitis (Infections and infestations) | 19 | 10 | 13 | 3
Pharyngitis (Infections and infestations) | 14 | 18 | 16 | 7
Upper respiratory tract infection (Infections and infestations) | 18 | 20 | 16 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.